CLINICAL TRIAL: NCT01226303
Title: Treatment Study for Children and Adolescents With Acute Promyelocitic Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICC APL STUDY 01
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-07

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard risk (Experimental): are defined as those patients with a WBC less than 10x10 9 /L at presentation
  Interventions: Drug: ATRA
- high risk (Active Comparator): are defined as those patients whose highest treatment WBC is equal to or greater than 10x10 9 /L at presentation
  Interventions: Drug: ATRA + IDA

INTERVENTIONS:
Drug: ATRA — see the protocol
  Arms: standard risk
Drug: ATRA + IDA — see the protocol
  Arms: high risk

SUMMARY:
This study is open to all patients with a diagnosis of acute promyelocytic leukemia (APL) who are PCR positive for the PML-RARα transcript or rarer retinoid sensitive subtypes (i.e. NPM-RAR-alpha, NuMA-RARalpha) and less than 21 years of age (for AIEOP, see appendix A).

DETAILED DESCRIPTION:
This study is open to all patients with a diagnosis of acute promyelocytic leukemia (APL) who are PCR positive for the PML-RARα transcript or rarer retinoid sensitive subtypes (i.e. NPM-RARalpha, NuMA-RARalpha) and less than 21 years of age (for AIEOP, see appendix A). APL is a rare disease with each national group recruiting small numbers of patients to their trials annually. Therefore this will be an international study expecting to recruit 60-70 patients per annum and a total of 300 patients in 5 years. The study aims to limit the use of anthracyclines and stratify treatment by risk group: standard risk - WBC <10 x 109/l : high risk - WBC ≥10 x 109/l. All-trans retinoic acid (ATRA) is included in all phases of therapy and intermediate dose Ara-C (IDARAC) is given during consolidation treatment. Following one induction course of treatment standard risk patients have 2 consolidation blocks whilst high risk patients have 3 consolidation blocks.

The PML-RARα transcript will be monitored throughout and standard risk patients with detectable minimal residual disease by real time quantitative reverse transcriptase polymerase chain reaction (RQ-PCR+) at the end of the second consolidation block will receive a third consolidation block identical to high risk patients. Patients who are RQ-PCR+ for PML-RARα after completion of the third block of consolidation therapy will be candidates for refractory/relapse treatment, but will remain on study. Refractory/relapsed patients who remain RQ-PCR+ for PML-RARα will be candidates for allogeneic bone marrow transplantation (allo-BMT), whilst those who become RQ-PCR- for PML-RARα will have individualised treatment with ongoing MRD monitoring.

These study guidelines are intended to describe a collaborative international study in APL in children and adolescents and to provide information about procedures for the entry, treatment and follow-up of patients. It is not intended that these guidelines be used as an aide-memoir or guide for the treatment of other patients. Every care has been taken in its drafting, but corrections and amendments may be necessary. Before entering patients into the study, clinicians must ensure that the study has received clearance from their Local Research Ethics Committee and any other necessary body.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of initial APL and subsequently confirmed to have PML-RARα, NPM1-RARα or NUMA-RARα fusion. Whilst this study is only for ATRA-sensitive APL, APL is a hematological emergency and ATRA should be commenced as soon as the diagnosis is suspected. Study entry should not wait until the diagnosis of APL has been confirmed molecularly or cytogenetically
* Less than 21 years of age at initial diagnosis (for AIEOP, see appendix A)
* Considered suitable for anthracycline-based chemotherapy
* Written informed consent available
* Females of childbearing age must have a negative pregnancy test and subsequently must attempt to avoid pregnancy

Exclusion Criteria:

* Patients with a clinical diagnosis of APL but subsequently found to have PLZF-RARα fusion or lacking PML-RARα, NPM-RARα or NuMA-RARα rearrangement should be withdrawn from the study and treated on an alternative protocol.
* Refractory/relapsed APL (the guidelines in this protocol for that subgroup are intended for patients treated from initial diagnosis according to this protocol)
* Concurrent active malignancy
* Pregnant or lactating
* Physician and patient/guardian think that intensive chemotherapy is not an appropriate treatment option
* Patients who have received alternative chemotherapy for 7 days or longer without ATRA for any reason (either APL not initially suspected or ATRA not available).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
• to conduct an international pediatric study for APL based on the GIMEMA-AIEOP/AIDA 93 protocol (the study from the Italian GIMEMA -AIEOP group which has produced the best results in children with APL to date), with optimal outcome and less toxicity | 5 years
  • to conduct an international pediatric study for APL based on the GIMEMA-AIEOP/AIDA 93 protocol (the study from the Italian GIMEMA -AIEOP group which has produced the best results in children with APL to date), with optimal outcome and less toxicity

SECONDARY OUTCOMES:
• To monitor cardiotoxicity by echocardiography | 5 years
  • To monitor cardiotoxicity by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Testi, Dr, Principal Investigator — Associazione Italiana Ematologia Oncologia Pediatrica
Locations (1):
- Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma, Italy

REFERENCES:
- See also: Italian association of Pediatric Hematology and Oncology — http://www.aieop.org